CLINICAL TRIAL: NCT06261307
Title: Language Development Deficits and Early Interactive Music Intervention - a Randomized Controlled Trial (BusyBaby)
Brief Title: Language Development Deficits and Early Interactive Music Intervention
Acronym: BusyBaby
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Folkhälsan Research Center (Unknown); Karolinska Institutet (Other); University of Turku (Other); University of Jyvaskyla (Other); Academy of Finland (Other)
Responsible Party: Principal Investigator, Paula Virtala, University researcher, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13462111
Record Dates: First submitted 2024-01-17; First posted 2024-02-15 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Dyslexia, Developmental; Language Development Disorders; Language Development
Keywords: Event-related potentials; Music intervention; Brain development; Speech processing
MeSH Terms: conditions — Dyslexia; Language Development Disorders

STUDY DESIGN:
Intervention Model Description: The experimental arm will receive music training and the control arm will receive circus training.
Who Masked: Participant, Outcomes Assessor
Masking Description: A dedicated member of the research team will be in charge of randomization of the participants to the two intervention arms, to ensure blindness of other team members. This member will not act as an outcomes assessor or a care provider.
  The study will be presented to the caregivers as evaluating the effect of hobbies on language development. Therefore, the caregivers should not consider either intervention as the control arm. Both arms are expected to be potentially beneficial for the children's development.
  Outcomes assessors will be unaware of the intervention arm and risk status (dyslexia risk vs no risk) of the children; caregivers will be reminded not to mention these to the researcher. Person in charge of randomization keeps track of violations of outcome assessor blindness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music intervention (Experimental): Groups: Children with (risk group, appr. 50%) or without (control group, appr. 50%) familial risk for dyslexia.
  In each arm, the children will follow the same training protocol consisting of weekly 0.5-1-hour training sessions for six months. Training sessions are organized at fixed times and locations in fixed groups of 5-10 parent-child dyads and an experienced instructor.
  The music intervention consists of social, structured and playful group sessions that involve joint singing, playing with musical instruments, moving to and listening to music. Based on the results of a previous intervention study by the investigators on the benefits of vocal music exposure on speech processing (Virtala et al., 2023), joint singing will be emphasized in the music intervention. The aims of the music intervention are to support caregiver-child interaction and the development of musical abilities.
  Interventions: Behavioral: Music intervention
- Circus intervention (Active Comparator): Groups: Children with (risk group, appr. 50%) or without (control group, appr. 50%) familial risk for dyslexia.
  In each arm, the children will follow the same training protocol consisting of weekly 0.5-1-hour training sessions for six months. Training sessions are organized at fixed times and locations in fixed groups of 5-10 parent-child dyads and an experienced instructor.
  The circus intervention consists of social, structured and playful group sessions that involve acrobatics and other age-appropriate motor exercises with the caregiver, and familiarizing with the art and equipment of circus and acrobatics. The aims of the circus intervention are to support caregiver-child interaction and the development of motor skills.
  Interventions: Behavioral: Circus intervention

INTERVENTIONS:
Behavioral: Music intervention — Group intervention focusing on musical activities
  Arms: Music intervention
Behavioral: Circus intervention — Group intervention focusing on acrobatics and circus activities
  Arms: Circus intervention

SUMMARY:
Investigators compare effects of 6-month music versus circus group interventions on language development in infants and toddlers with or without familial risk for dyslexia (anticipated total N=200). Effects of intervention timing, dyslexia risk and genetics, and social-emotional factors on the intervention outcomes are investigated.

DETAILED DESCRIPTION:
Infancy and early childhood lay the base for language and reading abilities, and this development can be compromised by heritable conditions such as the reading deficit developmental dyslexia. One of the earliest indices of language abilities is neural processing of native language speech, as it is associated both with familial risk for developmental language and reading deficits and with subsequent language and reading development. Previous work has shown that musical activities can promote auditory and language learning early on and even improve reading in dyslexic children. Large-scale randomized controlled trials are needed particularly in risk groups in order to give recommendations and design effective interventions to support language development and ameliorate later difficulties. The investigators will conduct such a trial to study the effects of a playful music training group compared to a similar circus training group on speech processing and language development in infancy and early childhood. It is investigated how these effects are moderated by familial risk for dyslexia and its genetic markers as well as timing of the intervention in relation to the children's age and developmental status. Investigators study how the expected social-emotional benefits of the interventions on the parent, child, and their interaction mediate the intervention effects on language. Approximately 8-12-month-old infants with confirmed parental dyslexia or without parental dyslexia will be randomized, using block randomization, to one of the two 6-month training groups, and outcome measures will be collected before and after the intervention and at follow-up ~1 year after the intervention has ended. The total anticipated sample size is 200, with approximately 100 infants in the music and circus interventions and within each intervention, approximately 50 infants with and 50 without parental dyslexia. Speech processing will be evaluated with speech-elicited auditory event-related potentials, and language skills and general development with standardized parental questionnaires and age-appropriate standardized tests. Social-emotional factors are evaluated with parental questionnaires. DNA samples are collected to study dyslexia genetics. The results can contribute to designing effective interventions for supporting language development in vulnerable groups early on.

ELIGIBILITY:
Inclusion Criteria:

* 8-12 months old at start of intervention (recruited between 0-11 months)
* Born healthy and at term (gestational age at least 37 weeks and birth weight at least 2500 g)
* Normal hearing at birth (evoked oto-acoustic emissions conducted to newborns routinely at the hospital)
* At least one caregiver living with the child is native speaker of Finnish and speaks Finnish to the child
* Risk group: At least one biological parent has developmental dyslexia according to a recent (<5 years) diagnostic statement by a health care professional or according to a dyslexia test at study enrollment; symptoms have started in childhood

Exclusion Criteria:

* Medication affecting the central nervous system
* Sensory deficits
* Serious health conditions
* No-risk group: Suspected dyslexia or developmental language disorder due to symptoms that have started in childhood in either of the biological parents; diagnosis of a developmental or language disorder (incl. dyslexia, developmental language disorder, attention-deficit/hyperactivity disorder ADHD, attention-deficit disorder ADD) or neurological disorder in either of the biological parents
* Risk group: Diagnosis of ADHD, ADD, or other not-language-related developmental disorder in either of the biological parents; in the dyslexic parent, brain trauma in childhood that may indicate a non-heritable cause for the reading deficit or individualized school curriculum that may indicate broader developmental deficits.

Ages: 8 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Infant-Toddler Checklist (ITC) | At baseline and at 6 months (post intervention)
  Total and sub-scale scores in the parental standardized questionnaire on prelinguistic skills: Infant-Toddler Checklist (ITC) in the Communication and Symbolic Behavior Scales Developmental Profile (Wetherby and Prizant, 2002; in Finnish: Laakso et al., 2011). Range of scores is 0-57 for the Total score, 0-26 for the Social subscale, 0-14 for the Speech subscale, and 0-17 for the Symbolic subscale, higher scores reflecting better prelinguistic skills.
MacArthur-Bates Communicative Development Inventory (MCDI) 8-16mo | At baseline and at 6 months (post intervention)
  Size of receptive and expressive vocabulary (amount of words out of a total of 380 words for each), and total score in the "gestures" scale (0-66, higher score reflecting better skills) in a parental standardized questionnaire on early language skills: the MacArthur-Bates Communicative Development Inventory (MCDI; Fenson et al., 1991; in Finnish: Lyytinen, 1999)
Mismatch response (MMR) speech, amplitude | At baseline and at 6 months (post intervention)
  Amplitude (in microvolts) of mismatch responses to speech sound deviants in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Mismatch response (MMR) speech, latency | At baseline and at 6 months (post intervention)
  Peak latency (in milliseconds) of mismatch responses to speech sound deviants in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Mismatch response (MMR) speech, laterality | At baseline and at 6 months (post intervention)
  Hemispheric lateralization (indicated with a laterality index, where range is from -1 to +1 with more positive values indicating a more left-lateralized response) of mismatch responses to speech sound deviants in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest at left and right hemisphere
Obligatory event-related potential (ERP) speech, amplitude | At baseline and at 6 months (post intervention)
  Amplitude (in microvolts) of obligatory event-related potentials (ERPs) to repeating speech sounds in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Obligatory event-related potential (ERP) speech, latency | At baseline and at 6 months (post intervention)
  Peak latency (in milliseconds) of obligatory event-related potentials (ERPs) to repeating speech sounds in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Obligatory event-related potential (ERP) speech, laterality | At baseline and at 6 months (post intervention)
  Hemispheric lateralization (indicated with a laterality index, where range is from -1 to +1 with more positive values indicating a more left-lateralized response) of obligatory event-related potentials (ERPs) to repeating speech sounds in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest at left and right hemisphere

SECONDARY OUTCOMES:
Infant-Toddler Checklist (ITC) follow-up | At 1-year follow-up (1.5 years from baseline)
  Total and sub-scale scores in the standardized parental questionnaire on prelinguistic skills: Infant-Toddler Checklist (ITC) in the Communication and Symbolic Behavior Scales Developmental Profile (Wetherby and Prizant, 2002; in Finnish: Laakso et al., 2011). Range of scores is 0-57 for the Total score, 0-26 for the Social subscale, 0-14 for the Speech subscale, and 0-17 for the Symbolic subscale, higher scores reflecting better prelinguistic skills.
MacArthur-Bates Communicative Development Inventory (MCDI) 16-30mo follow-up | At 1-year follow-up (1.5 years from baseline)
  Size of expressive vocabulary (amount of words out of a total of 595 words) and mean length of utterance (mean number of morphemes in the three longest utterances used by the child) in a parental standardized questionnaire on early language skills: the MacArthur-Bates Communicative Development Inventory (MCDI; Fenson et al., 1991; in Finnish: Lyytinen, 1999)
Mismatch response (MMR) speech, amplitude follow-up | At 1-year follow-up (1.5 years from baseline)
  Amplitude (in milliseconds) of mismatch responses to speech sound deviants in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Mismatch response (MMR) speech, latency follow-up | At 1-year follow-up (1.5 years from baseline)
  Peak latency (in milliseconds) of mismatch responses to speech sound deviants in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Mismatch response (MMR) speech, laterality follow-up | At 1-year follow-up (1.5 years from baseline)
  Hemispheric lateralization (indicated with a laterality index, where range is from -1 to +1 with more positive values indicating a more left-lateralized response) of mismatch responses to speech sound deviants in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest at left and right hemisphere
Obligatory event-related potential (ERP) speech, amplitude follow-up | At 1-year follow-up (1.5 years from baseline)
  Amplitude (in milliseconds) of obligatory event-related potentials (ERPs) to repeating speech sounds in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Obligatory event-related potential (ERP) speech, latency follow-up | At 1-year follow-up (1.5 years from baseline)
  Peak latency (in milliseconds) of obligatory event-related potentials (ERPs) to repeating speech sounds in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Obligatory event-related potential (ERP) speech, laterality follow-up | At 1-year follow-up (1.5 years from baseline)
  Hemispheric lateralization (indicated with a laterality index, where range is from -1 to +1 with more positive values indicating a more left-lateralized response) of obligatory event-related potentials (ERPs) to repeating speech sounds in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest at left and right hemisphere
Reynell Developmental Language Scales III (RDLS-III) | At 6 months (post intervention) and at 1-year follow-up (1.5 years from baseline)
  Expressive and Comprehension Scale scores in the standardized language test battery Reynell Developmental Language Scales III (Reynell and Huntley, 2001). The range of scores is 0-62 for both scales, higher scores reflecting better language abilities.
Infant Behavior Questionnaire Revised short form (IBQ-R-sf) | At baseline
  Factor scores in a parental standardized questionnaire on infant temperament at baseline: Infant Behavior Questionnaire Revised short form (IBQ-R, Putnam et al. 2014). The range of scores, with higher scores reflecting stronger trait, for the three factors are, for Negative affectivity, 1-6.25, for Surgency/Extraversion, 1-6.66, and for Orienting/Regulation/Effortful control, 1-6.5.
Early Childhood Behavior Questionnaire short form (ECBQ-sf) | At 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Factor scores in a parental standardized questionnaire on early childhood temperament at six months and 1.5 years from baseline: Early Childhood Behavior Questionnaire short form (ECBQ-sf, Putnam et al. 2010). The range of scores, with higher scores reflecting stronger trait, for the three factors are, for Negative affectivity, 1-6, for Surgency/Extraversion, 1-5.4, and for Orienting/Regulation/Effortful control, 1-6.4. The questionnaire is continuation to the Infant Behavior Questionnaire Revised short form (IBQ-R-sf), allowing the analysis of change in factor scores from baseline.
Parenting Stress Index Short Form (PSI-sf) | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Factor and total stress scores in a parental standardized questionnaire on parental well-being and stress and interaction with child: Parenting Stress Index Short Form (PSI-sf, Abidin, 1995). The range of scores is 12-60 for the three factors Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child, and sum of these (36-180) for the Total score, with higher scores indicating more challenges (poorer parental well-being, more stress, and more dysfunctional interaction with the child).
Brief Infant-Toddler Social Emotional Assessment (BITSEA) | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Problem and Competence scores in a parental standardized questionnaire on social-emotional/behavioral problems and delays in social-emotional competence: Brief Infant-Toddler Social Emotional Assessment (BITSEA, Briggs-Gowan et al. 2004). The range for the Problem scores is 0-62, higher scores reflecting more problems in social-emotional skills or behavior. The range for the Competence scores is 0-22, higher scores reflecting better social-emotional competence. Both the scores and their percentile rankings (dependent on age and gender of the child, lower percentile always indicating worse performance) are analyzed.

OTHER OUTCOMES:
Parental dyslexia status (dyslexia - no dyslexia) | At enrollment to the study (before the children are accepted to the study and randomized)
  Parental dyslexia status confirmed with a recent (< 5 years) clinical statement or a test battery including a clinical interview and a standardized questionnaire, described, e.g. in Kujala et al. (2021). Parental dyslexia is an inclusion criterion for the risk group participants, and it will be evaluated from all parents who suspect that they have dyslexia.
Allele groupings for dyslexia susceptibility genes | At baseline
  Allele groupings in single nucleotide polymorphisms (SNPs) of susceptibility genes associated with language, reading, and developmental dyslexia, analyzed from DNA samples and used for forming subgroups to study associations to Outcome measures 1-17. After data collection ends for the outcome measures, 5-10 most relevant SNPs are chosen according to the most recent research literature.
Gross and fine motor development | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Ages of reaching basic milestones in gross motor development and fine motor development, as reported by parents in a background questionnaire
Bayley Scales III Motor scale | At 6 months (post-intervention) and at 1-year follow-up (1.5 years from baseline)
  Fine and gross motor development of the child as evaluated with the Motor scale of the standardized Bayley Scales III battery (Bayley, 2006).The range of scores for the Fine motor development scale is 0-66 and for the Gross motor development scale, 0-72, higher scores reflecting better motor abilities.
Mismatch response (MMR) music, amplitude | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Amplitude (in microvolts) of mismatch responses to auditory deviants in a musical oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Mismatch response (MMR) music, latency | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Peak latency (in milliseconds) of mismatch responses to auditory deviants in a musical oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Mismatch response (MMR) music, laterality | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Hemispheric lateralization (indicated with a laterality index, where range is from -1 to +1 with more positive values indicating a more left-lateralized response) of mismatch responses to auditory deviants in a musical oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Obligatory event-related potential (ERP) music, amplitude | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Amplitude (in microvolts) of obligatory event-related potentials (ERPs) to repeating musical stimuli in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Obligatory event-related potential (ERP) music, latency | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Peak latency (in milliseconds) of obligatory event-related potentials (ERPs) to repeating musical stimuli in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest
Obligatory event-related potential (ERP) music, laterality | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Hemispheric lateralization (indicated with a laterality index, where range is from -1 to +1 with more positive values indicating a more left-lateralized response) of obligatory event-related potentials (ERPs) to repeating musical stimuli in an oddball paradigm recorded with electroencephalogram (EEG) from a fronto-central region-of-interest at left and right hemisphere
Music test scores (three parts of MMBB-MB) | At 1-year follow-up (1.5 years from baseline)
  A custom-made musicality test battery, i.e., the Music, Mind, Body, and Brain Music Battery (MMBB-MB) measures core domains of music cognition. The children (with the help of their parents, according to their age-appropriate abilities) are asked 1) to tap with their finger in unpaced (spontaneous) and paced (to metronome and music) conditions, 2) to perform whole-body movements in unpaced and paced conditions, and 3) to sing along models or spontaneously single tones, tone sequences, and a familiar song.
Music-related activities | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Frequency and intensity of child's music-related activities as reported by parents in a background questionnaire (incl. joint singing, dancing, moving to music and playing instruments at home, music listening and exposure to music at home, music-related hobbies)
Musical background of parents | At baseline
  Parents' musical background (incl. preferences, training, and listening habits) self-reported in a background questionnaire
Home literacy | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Quality of home literacy environment (incl. amount of reading in parents, amount of reading aloud to the child, amount of children's and adults' books at home, frequency of library visits, and audio book listening) as reported by parents in a background questionnaire
Multilingualism | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  The degree of multilingualism of the child and their environment (incl. native languages of family members and languages spoken to the child at home, at daycare, and at other environments) as reported by parents in a background questionnaire
Screen time | At baseline, 6 months (post-intervention), and 1-year follow-up (1.5 years from baseline)
  Total weekly screen time of the child in hours as reported by parents in a background questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Paula Virtala, PhD, Principal Investigator — University of Helsinki
Locations (1):
- University of Helsinki, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paula V, Vesa P, Anastasia G, Anja T, Laurel J T, Teija K. Beneficial effects of a music listening intervention on neural speech processing in 0-28-month-old children at risk for dyslexia. Dev Sci. 2023 Sep;26(5):e13426. doi: 10.1111/desc.13426. Epub 2023 Jun 23. PMID 37350469
- [Background] Kujala T, Sihvonen AJ, Thiede A, Palo-Oja P, Virtala P, Numminen J, Laasonen M. Voxel and surface based whole brain analysis shows reading skill associated grey matter abnormalities in dyslexia. Sci Rep. 2021 May 25;11(1):10862. doi: 10.1038/s41598-021-89317-x. PMID 34035329
- [Derived] Virtala P, Aquilino B, Nie P, Navarrete-Arroyo S, Stolt S, Leutonen K, Lauronen M, Kujala T. Language development deficits and early interactive music intervention (BusyBaby): protocol description of a double-blind randomized controlled trial on the effectiveness of music on language development in infancy. Front Psychol. 2026 Jan 5;16:1699558. doi: 10.3389/fpsyg.2025.1699558. eCollection 2025. PMID 41561604